CLINICAL TRIAL: NCT04514393
Title: Phase II Study of Combination Treatment of Methotrexate, Ibrutinib, and Temozolomide (MIT Regimen) in Patients With Newly Diagnosed Primary CNS Lymphoma
Brief Title: Ibrutinib With Methotrexate and Temozolomide for Patients With Newly Diagnosed Primary CNS Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huiqiang Huang (Other)
Collaborators: Guangdong 999 Brain Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Xian-Janssen Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIT
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Primary Central Nervous System Lymphoma; PCNSL; Non Hodgkin Lymphoma
Keywords: PCNSL; Newly Diagnosed
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Methotrexate; ibrutinib; Temozolomide

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- methotrexate, ibrutinib, and temozolomide (MIT regimen) (Experimental): Methotrexate will be given on day 1 of each 28-day cycle；Ibrutinib will be given day 1-28 of each 28-day cycle; Temozolomide will be given day 1-5 of each 28-day cycle. Methotrexate and Temozolomide are given for up to 4 cycles; Ibrutinib is continued until disease progression, intolerable toxicity, or death.
  Interventions: Drug: Methotrexate; Drug: Ibrutinib; Drug: Temozolomide

INTERVENTIONS:
Drug: Methotrexate — Intravenous methotrexate at 3.5g/m2 (standard hydration/leucovorin support) will be given on day 1 of all cycles，for up to 4 cycles.
  Other Names: MTX
Drug: Ibrutinib — Oral ibrutinib will be given at a dose of 560 mg daily and will be continued daily after completion of methotrexate and temozolomide.Ibrutinib is continued until disease progression, intolerable toxicity or death.
  Other Names: Imbruvica
Drug: Temozolomide — Oral temozolomide will be given at 150mg/m2 from day1 to day 5 every 4 of all cycles，for up to 4 cycles.
  Other Names: TMZ

SUMMARY:
The purpose of the study is to test the efficacy and tolerability of a combination treatment of methotrexate, ibrutinib, and temozolomide (MIT regimen) in treating patients who have newly-diagnosed primary CNS lymphoma.

DETAILED DESCRIPTION:
Primary central nervous system lymphoma (PCNSL) is a rare and aggressive extranodal Non-Hodgkin Lymphoma. Induction treatment of PCNSL in most reported single-arm or randomized trials includes high-dose methotrexate (HD-MTX)-based therapy, temozolomide, with or without cytarabine and the anti-CD20 antibody rituximab. A better combination remains undefined. Treatment is associated with considerable morbidity and disease recurrences with a 5-year survival of approximately 40%.

The BTK inhibitor ibrutinib has shown antitumor activity in patients with recurrent or refractory PCNSL. However, tumor responses to single-agent ibrutinib in CNS lymphoma are often incomplete or transient. Efficacy and safety of ibrutinib in combination with cytotoxic agents are worth to be discovered. Grommes et al.have shown ibrutinib in combination with methotrexate and rituximab are safe and shows promising activity in recurrent/refractory CNS lymphoma. In comparison to their prior study with single-agent ibrutinib, the radiographic response of r/r PCNSL was higher with the ibrutinib/HD-MTX/rituximab combination regimen and PFS was longer with the combination therapy. The study has shown that ibrutinib combined with chemotherapy were superior to ibrutinib single agent and overcome the transient effect of ibrutinib in relapsed PCNSL. However, there are some limitations in interpreting Grommes' study results, especially the heterogeneous patient population with inclusion of both PCNSL and SCNSL. Most recently, the role of rituximab in PCNSL has become clearly. In the HOVON 105/ALLG NHL 24 study, the addition of rituximab to a methotrexate-based regimen did not demonstrate a significant benefit on clinical outcome. We therefore initiate this study aim to evaluate the activity and safety of ibrutinib in combination with Methotrexate and temozolomide (MIT regimen) in newly diagnosed PCNSL patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and woman who are 18 to 70 years of age on the day of consenting to the study.
* Histologically documented PCNSL
* ECOG performance status ≤ 2.
* Life expectancy of > 3 months (in the opinion of the investigator).
* Adequate bone marrow and organ function shown by:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelets ≥ 75 x 10^9/L and no platelet transfusion within the past 14 days prior to study registration
  * Hemoglobin (Hgb) ≥ 8 g/dL and no red blood cell (RBC) transfusion within the past 14 days prior to study registration
  * International Normalized Ratio (INR) ≤ 1.5 and PTT (aPTT) ≤ 1.5 times the upper limit of normal
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal
  * Serum bilirubin ≤ 1.5 times the upper limit of normal; or total bilirubin ≤ 3 times the upper limit of normal with direct bilirubin within the normal range in patients with well documented Gilbert Syndrome
  * Serum creatinine ≤ 2 times the upper limit of normal
  * Lipase ≤ 1.5 x upper limit of normal
* Women of childbearing potential (WOCBP) and men must agree to use effective contraception when sexually active. This applies for the time period between signing of the informed consent form and 30 days (for WOCBP) and 90 days (for men) after the last administration of study treatment. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include but are not limited to hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for continuous 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy.

  * The investigator or a designated associate is requested to advise the patient how to achieve highly effective birth control (failure rate of less than 1%), e.g. intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner and sexual abstinence
  * The use of condoms by male patients is required unless the female partner is permanently sterile. Female subjects of childbearing potential must have a negative plasma pregnancy test upon study entry
* Must be able to tolerate MRI/CT scans
* Must be able to tolerate lumbar puncture and/or Ommaya taps
* Able to submit up to 20 unstained formalin-fixed, paraffin-embedded (FFPE) slides from the initial or most recent tissue diagnosis for correlative studies

Exclusion Criteria:

Patients eligible for this study must NOT MEET ANY of the following criteria:

• Active concurrent malignancy requiring active therapy

Excluded medical conditions:

* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure (New York Heart Association > Class 2), unstable angina, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Uncontrolled hypertension despite optimal medical management (per investigators assessment)
* Patient has poorly controlled diabetes mellitus with a glycosylated hemoglobin >8% or poorly controlled steroid-induced diabetes mellitus with a glycosylated hemoglobin of >8%
* Patient is known to have an uncontrolled active systemic infection (>CTCAE grade 2) and recent infection requiring intravenous anti-infective treatment that was completed ≤14 days before the first dose of study drug
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident, deep vein thrombosis or pulmonary embolism within 3 months before the start of study treatment
* Non-healing wound, ulcer or bone fracture
* Known bleeding diathesis (eg, von Willebrands disease) or hemophilia
* Known history of infection with human immunodeficiency virus (HIV) or active stage of infection with hepatitis C virus (HCV) or hepatitis B virus (HBV) as determined by serologic tests, or any uncontrolled active systemic infection
* Patient underwent major systemic surgery ≤ 2 weeks prior to starting the trial treatment or who has not recovered from the side effects of such surgery, or who plan to have surgery within 2 weeks of the first dose of the study drug
* Unable to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction
* Any life-threatening illness, medical condition including uncontrolled diabetes mellitus (DM), uncontrolled hypertension or organ system dysfunction that, in the opinion of the investigator, could compromise the subjects safety or put the study outcomes at undue risk
* Lactating or pregnant

Excluded previous Therapies and medications:

* Concurrent use of warfarin or other vitamin K antagonists (need to be stopped 7 days prior to starting on trial drug)
* Concurrent use of a strong cytochrome P450 (CYP) 3A4/5 inhibitor and inducers (need to be stopped 2 weeks prior to starting on trial drug)
* Enzyme-inducing antiepileptic drugs (EIAED) need to be discontinued and switched to a non-EIAED 2 weeks prior to starting on trial drug)
* Patient requires more than 4 mg of dexamethasone daily or the equivalent
* Patient is using systemic immunosuppressant therapy, including cyclosporine A, tacrolimus, sirolimus, and other such medications, or chronic administration of > 5 mg/day or prednisone or the equivalent. Participants must be off of immunosuppressant therapy for at least 28 days prior to the first dose of the study drug
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc., or chronic administration of > 5 mg/day of prednisone) within 28 days of the first dose of study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
the overall response (complete response + partial response)，Investigator-Assessed | up to 24 months
  The overall response rate (ORR) including complete response (CR), unconfirmed complete (CRu) and partial response (PR) according to the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG)
the toxicity profile of the ibrutinib/MTX/ temozolomide combination therapy | up to 24 months
  All subjects who received at least one dose of MIT will be included in the safety analysis. Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0. Treatment-emergent adverse events (TEAEs) will be summarised and tabulated according to the primary system organ class and preferred term. Type, incidence, severity, and seriousness of adverse events (AEs) including physical examination, safety laboratory parameters, vital signs, and so on will be analyzed.

SECONDARY OUTCOMES:
Complete response (CR) rate | up to 24 months
  The CR rate is defined as the proportion of patients who achieve complete remission(CR)/unconfirmed complete (CRu) based on the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG).
Duration of response（DOR） | up to 24 months
  Duration of response is defined as the time from the date of first occurrence of CR or PR to the date of the first documented PD or death due to any cause.
Progression-free survival (PFS) | 1 year and 2 years
  1 year and 2 years PFS rate.Disease progression was based on the 2005 Response Criteria of the International Primary CNS Lymphoma Collaborative Group (IPCG)
overall survival (OS) | 1 year and 2 years
  1-year and 2-year OS rates.

OTHER OUTCOMES:
Describe the tumor mutation profile by NGS | up to 24 months
  DNA from tumor tissue and CSF will be sequencing by next generation sequencing (NGS).Identify the PNCSL-related variants and gene expression alterations by NGS.
Relationship between prognostic and gene mutation in patients with PCNSL | up to 24 months
  Will be correlated with treatment response, mutational analysis using next-generation sequencing, and characterization of aberrant gene expression in PCNSL samples

CONTACTS AND LOCATIONS:
Overall Officials: Huiqiang Huang, Professor, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Department of Hematology Nanfang Hospital, The Southern Medical University, Guandong, Guangdong
  - Department of Medical Oncology, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong 999 Brain Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No